CLINICAL TRIAL: NCT06636968
Title: A Real-world Study to Evaluate the Effectiveness of Intravascular Lithotripsy in Moderate to Severe Calcification Lesion of Lower Extremity Femoropopliteal Artery
Acronym: STRIKE
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: RenJi Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Huashan Hospital (Other); Dongfang Hospital Affiliated to Tongji University (Other); Xuanwu Hospital, Beijing (Other); Qingdao Haici Hospital (Other); Second Affiliated Hospital of Soochow University (Other); First Affiliated Hospital of Fujian Medical University (Other); Quanzhou First Hospital (Other); The Second Affiliated Hospital of Hainan Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); First Hospital of China Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: The STRIKE study; B2024-270 (Other: Zhongshan Hospital)
Record Dates: First submitted 2024-09-23; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease
Keywords: calcification lesion; intravascular lithotripsy; lower-extremity arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Vascular calcification is prevalent in patients with Peripheral artery disease (PAD), especially those with combined diabetes or chronic kidney disease. Severe calcification predicts poor prognosis and is independently associated with increased risk of cardiovascular death and morbidity. Calcification may also affect the outcome of endovascular therapy, leading to unsatisfactory vasodilation, and increase the risk of vascular complications (including restenosis) and dissection, perforation, and distal embolization. At present, according to the degree of calcification and the scope of the lesion, it can be divided into light, medium and severe three grades. Neither high pressure balloon nor atherectomy can significantly improve severe calcification. The efficacy of these treatments has also not been tested in multicenter, real-world studies. Shockwave balloon has been widely used in the clinical treatment of severe calcification due to its characteristics of significantly destroying the calcification structure, reducing the damage of vascular intima, and thus reducing postoperative complications. The currently published Disrupt PAD III Trial (NCT02923193) in calcified lesions showed shock wave balloon versus balloon expansion alone in a randomized controlled trial (RCT). The residual stenosis rate was lower (66.4% vs. 51.9%; p = 0.02), the incidence of fluid limiting intersections was low (1.4% vs. 6.8%; p = 0.03), the rate of post-expansion and recovery support was also low (5.2% vs. 17.0%; p = 0.001); (4.6% vs. 18.3%; p < 0.001). The shock wave balloon has been approved by the China Food and Drug Administration for the intracavitary treatment of severe femoral popliteal artery calcification. Due to its short market-time, it is currently only used in large vascular surgery centers. On this basis, investigators propose whether can set up a real-world study of shock wave balloon in the treatment of moderate and severe calcification, in order to explore the real efficacy of shock wave balloon in the treatment of moderate and severe calcification.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Rutherford scale: Grades 2-5.
* Moderate-severe calcification of lower extremity arteries (defined as calcification on both sides of the arteries, the length of the lesion greater than 5cm).
* The stenosis degree of the lesions was more than 70% confirmed by DSA, including chronic occlusive lesions.
* At least one sub-knee branch artery is patent (defined as a run-off score of 1 or less). • In-stent restenosis or restenosis with moderate to severe calcification.
* The stenosis degree of inflow blood vessel on the diseased side is less than 30% or the residual stenosis is less than 30% after first-stage treatment.
* Calcification lesions with thrombus can also be included in the group after the thrombus is completely cleared.
* Sign relevant informed consent.

Exclusion Criteria:

* Active infection of the affected limb.
* Patients with severe ischemia of the affected limb who are expected to undergo major amputation.
* The target blood vessels were artificial blood vessels or autologous vessels.
* Simple thrombosis lesion.
* Thromboangiitis obliterans, arteritis or connective tissue disease-based lesions.
* Inflow vessel stenosis is greater than 30% or residual stenosis is still greater than 30% after primary treatment.
* Allergic to contrast agent, heparin, anti-platelet therapy.
* Patients who are pregnant or lactating.
* Patients with cardiovascular and cerebrovascular events such as stroke or myocardial infarction within 3 months prior to enrollment.
* Patients who are currently in an ongoing interventional clinical study program.
* Patients who refuse to sign informed consent. •
* Patients who refuse to cooperate with long-term follow-up after surgery or who, for personal reasons, have difficulty communicating for quality of life assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) Age more than 18 years old; (2) Smoking, diabetes, hypertension, hyperlipidemia and other high risk factors; (3) Clinical manifestations of lower extremity arteriosclerosis obliterans; (4) The distal artery pulsation of the ischemic limb is weakened or disappeared (5)ABI≤0.9; (6) Color Doppler ultrasound, CT angiography (CTA), magnetic resonance angiography (MR angiography) and Digital subtraction angiography (Digital subtraction angiography) angiography, Imaging tests such as DSA showed the stenosis or occlusion of the corresponding arteries. (6)Moderate-severe calcification of lower extremity arteries (defined as calcification on both sides of the arteries, the length of the lesion greater than 5cm).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical Success rate | 7 Days
  Defined as a final residual stenosis of less than 30% without a significant dissection (grade ≥D)

SECONDARY OUTCOMES:
Bailout stent | 7 Days
  The rate of bailout stent implantation.
Composite MAEs and embolization | 1 month
  Composite end point of major amputation plus operation-associated arterial embolization.
operation-associated arterial embolization | 7 Days
  Perioperative operation-associated arterial embolization
Dissection severity | 1 Day
  Dissection after major procedure
Dissection severity-last | 1 Day
  Dissection after last procesure
Major amputation | 1 year
  Major amputation rate in different frame
Primary patency | 1 year
  Primary patency in different frame
Freedom from TLR | 1 year
  Freedom from TLR in different frame
Rutherford category | 1 year
  Rutherford grading improvement score after surgery（Rutherford Classification,0-6, higher scores mean a worse outcome）
quality of life score | 1 year
  Postoperative quality of life score(15-items quality of recovery scale after, 0-150, higher scores mean a better outcome)
Indicators of health economics | 7 Days
  Cumulative hospitalization costs associated with target lesions and costs associated with endovascular therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia Del Blanco B, Seidelberger B, Iniguez A, Gomez-Recio M, Masotti M, Velazquez MT, Sanchis J, Garcia-Touchard A, Zueco J, Bethencourt A, Melgares R, Cequier A, Dominguez A, Mainar V, Lopez-Minguez JR, Moreu J, Marti V, Moreno R, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS V Study Investigators, under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology. A randomized comparison of drug-eluting balloon versus everolimus-eluting stent in patients with bare-metal stent-in-stent restenosis: the RIBS V Clinical Trial (Restenosis Intra-stent of Bare Metal Stents: paclitaxel-eluting balloon vs. everolimus-eluting stent). J Am Coll Cardiol. 2014 Apr 15;63(14):1378-86. doi: 10.1016/j.jacc.2013.12.006. Epub 2014 Jan 8. PMID 24412457
- [Background] Werk M, Albrecht T, Meyer DR, Ahmed MN, Behne A, Dietz U, Eschenbach G, Hartmann H, Lange C, Schnorr B, Stiepani H, Zoccai GB, Hanninen EL. Paclitaxel-coated balloons reduce restenosis after femoro-popliteal angioplasty: evidence from the randomized PACIFIER trial. Circ Cardiovasc Interv. 2012 Dec;5(6):831-40. doi: 10.1161/CIRCINTERVENTIONS.112.971630. Epub 2012 Nov 27. PMID 23192918
- [Background] Liistro F, Porto I, Angioli P, Grotti S, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for below the knee angioplasty evaluation (DEBATE-BTK): a randomized trial in diabetic patients with critical limb ischemia. Circulation. 2013 Aug 6;128(6):615-21. doi: 10.1161/CIRCULATIONAHA.113.001811. PMID 23797811
- [Background] Jia X, Zhang J, Zhuang B, Fu W, Wu D, Wang F, Zhao Y, Guo P, Bi W, Wang S, Guo W. Acotec Drug-Coated Balloon Catheter: Randomized, Multicenter, Controlled Clinical Study in Femoropopliteal Arteries: Evidence From the AcoArt I Trial. JACC Cardiovasc Interv. 2016 Sep 26;9(18):1941-9. doi: 10.1016/j.jcin.2016.06.055. PMID 27659572
- [Background] Tarricone A, Ali Z, Rajamanickam A, Gujja K, Kapur V, Purushothaman KR, Purushothaman M, Vasquez M, Zalewski A, Parides M, Overbey J, Wiley J, Krishnan P. Histopathological Evidence of Adventitial or Medial Injury Is a Strong Predictor of Restenosis During Directional Atherectomy for Peripheral Artery Disease. J Endovasc Ther. 2015 Oct;22(5):712-5. doi: 10.1177/1526602815597683. Epub 2015 Jul 24. PMID 26208657
- [Background] Iida O, Takahara M, Soga Y, Hirano K, Yamauchi Y, Zen K, Yokoi H, Uematsu M; ZEPHYR investigators. Incidence and its characteristics of repetition of reintervention after drug-eluting stent implantation for femoropopliteal lesion. J Vasc Surg. 2016 Dec;64(6):1691-1695.e1. doi: 10.1016/j.jvs.2016.05.074. Epub 2016 Aug 27. PMID 27575807
- [Background] Zeller T, Dake MD, Tepe G, Brechtel K, Noory E, Beschorner U, Kultgen PL, Rastan A. Treatment of femoropopliteal in-stent restenosis with paclitaxel-eluting stents. JACC Cardiovasc Interv. 2013 Mar;6(3):274-81. doi: 10.1016/j.jcin.2012.12.118. PMID 23517839
- [Background] Dominguez A 3rd, Bahadorani J, Reeves R, Mahmud E, Patel M. Endovascular therapy for critical limb ischemia. Expert Rev Cardiovasc Ther. 2015 Apr;13(4):429-44. doi: 10.1586/14779072.2015.1019472. Epub 2015 Mar 2. PMID 25728744
- [Background] Xu Z, Ran X. Diabetic foot care in China: challenges and strategy. Lancet Diabetes Endocrinol. 2016 Apr;4(4):297-8. doi: 10.1016/S2213-8587(16)00051-6. No abstract available. PMID 27016321
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Result] Tepe G, Brodmann M, Werner M, Bachinsky W, Holden A, Zeller T, Mangalmurti S, Nolte-Ernsting C, Bertolet B, Scheinert D, Gray WA; Disrupt PAD III Investigators. Intravascular Lithotripsy for Peripheral Artery Calcification: 30-Day Outcomes From the Randomized Disrupt PAD III Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1352-1361. doi: 10.1016/j.jcin.2021.04.010. PMID 34167675